CLINICAL TRIAL: NCT01474395
Title: NMDA and Cognitive Remediation in Schizophrenia
Brief Title: N-methyl-D-aspartic Acid (NMDA) and Cognitive Remediation in Schizophrenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1115-00
Record Dates: First submitted 2011-10-06; First posted 2011-11-18 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2011-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; cognitive remediation; NMDA
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-serine 60 mg/kg (Experimental): double blind dose of d-serine
  Interventions: Drug: D-serine; Behavioral: Sensory Based remediation paradigm
- Placebo D-serine (Placebo Comparator)
  Interventions: Drug: placebo; Behavioral: Sensory Based remediation paradigm

INTERVENTIONS:
Drug: D-serine — Subjects will then undergo three treatment visits. Each visit will begin with a pre treatment MMN/visual motion paradigm. Subjects will then receive DSR (60 mg/kg) or placebo and begin a one-hour SBR intervention. SBR will begin approximately 30 minutes after drug administration, to coincide with peak serum DSR level. Finally, to evaluate the effects of SBR and NMDA treatment on neurophysiology, subjects will complete a post treatment ERP paradigm. Treatment days will be separated by 1 week to reduce carryover effect. To increase power, each subject will undergo two DSR treatment days and 1 placebo day, with the placebo day selected randomly from among the three treatment days, in counter balanced order. Treatment assignment (drug and SBR) will be double blinded. Follow-up cognitive and safety measures will also be completed on the final treatment day.
  Arms: D-serine 60 mg/kg
Drug: placebo — Subjects will then undergo three treatment visits. Each visit will begin with a pre treatment MMN/visual motion paradigm. Subjects will then receive DSR (60 mg/kg) or placebo and begin a one-hour SBR intervention. SBR will begin approximately 30 minutes after drug administration, to coincide with peak serum DSR level. Finally, to evaluate the effects of SBR and NMDA treatment on neurophysiology, subjects will complete a post treatment ERP paradigm. Treatment days will be separated by 1 week to reduce carryover effect. To increase power, each subject will undergo two DSR treatment days and 1 placebo day, with the placebo day selected randomly from among the three treatment days, in counter balanced order. Treatment assignment (drug and SBR) will be double blinded. Follow-up cognitive and safety measures will also be completed on the final treatment day.
  Arms: Placebo D-serine
Behavioral: Sensory Based remediation paradigm — Every subject will receive sensory based remediation on each treatment visit: Three 80-tone pair blocks will be used per session (~1 hour with breaks). To minimize practice effects, we will use a different base tone for each treatment day (e.g. 500, 1000, and 2000 Hz), also in a randomized counter-balanced order. To assess the improvement over a treatment day, we will record the ratio of the frequencies in all tone pairs. To correct this non-normal distribution we take the natural log of each of these ratios to determine the tone matching threshold.

SUMMARY:
Persistent neurocognitive deficits are a major cause of severe disability and impaired long-term psychosocial outcome in schizophrenia (SZ). In particular, within the auditory system, early deficits such as the behavioral and neurophysiological ability to match tones that vary in pitch correlate with impairments in auditory emotion recognition (affective prosody) and general functioning, suggesting that interventions aimed at remediating sensory-level dysfunction may lead to significant improvement in higher order cognitive/emotion processes. Efforts to ameliorate cognitive deficits in schizophrenia utilize either pharmacological agents or behavioral treatments such as cognitive remediation, which generally focus on higher order processes, and not on the early sensory processing which may be key to functioning.

Numerous pharmacological agents have been proposed, but accumulating evidence suggests that dysfunction of the N-methyl-D-aspartic acid (NMDA) receptor may be one of the root causes of schizophrenia, including sensory and cognitive impairments, suggesting that an NMDA based treatment may be efficacious in reversing these deficits. D-Cycloserine, a synthetic partial NMDA agonist has been used in anxiety disorders to augment learning in cognitive remediation. Because of a tendency to act as an NMDA antagonist at higher doses D-cycloserine is not effective in schizophrenia. In contrast, D-serine (DSR), is a full agonist, and is therefore more ideal for enhancing NMDA function and cognitive remediation. While previous use of DSR was limited by safety concerns in rodents,the investigators have shown that it can safely be used at doses of 60 mg/kg and, moreover, demonstrates converging improvement in symptomatic, cognitive and sensory-based measures in schizophrenia. Evidence also suggests that NMDA receptor dysfunction in schizophrenia may be relative, rather than absolute, suggesting that the enhanced practice of a cognitive remediation paradigm might be able to overcome reduced plasticity and treat cognitive dysfunction.

This project will be the first to combine the NMDA based and sensory-based cognitive remediation (SBR) approaches, and will utilize not only DSR, but also a tone matching SBR paradigm has been shown to enhance learning in healthy controls, as well as a paradigm designed to augment visual motion detection. This study will pilot these interventions in a double-blind, placebo-controlled, randomized crossover design that will use neurophysiology together with cognitive tests to explore the effects on brain activity and cognitive function in 16 patients with schizophrenia or schizoaffective disorder. The investigators hypothesize that DSR+SBR will lead to improvement. Subjects will have an initial visit to establish baseline performance on cognitive tasks before returning for 3 visits when they will receive blinded study medication [60 mg/kg of DSR (2 days) or placebo (1 day)] in a randomized order. The procedures on the treatment days will include the SBR paradigm and pre/post neurophysiological measurements. Primary outcomes are improvements in neurophysiologic and behavioral sensory processing. The main goal is to establish the preliminary efficacy to use in a follow-up multi-dose study utilizing a multiple session SBR R01 application.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years old, IQ≥85 and estimated Glomerular Filtration Rate (GFR) < or =60. All oral and depot antipsychotics (with the exception of clozapine) are allowable.
* Patients must be on their antipsychotic medication for 1 month and stable on dose of antipsychotic and adjunctive medications for 2 weeks prior to study entry.

Exclusion Criteria:

* Include a history of neurological visual or hearing impairment, active suicidal ideation on the Calgary Depression Scale (CDS), current alcohol or drug abuse (<1 month) or substance dependence (<4 months).
* All women of child-bearing potential must have a negative serum pregnancy test at the baseline visit.
* We require an IQ of greater or equal to 85 to ensure that subjects will have a capacity to learn.
* In our cross-sectional studies, we have observed an IQ greater than 85 in over 90% of candidates, suggesting that this is not an overly restrictive criterion.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Tone Matching threshold | 3 weeks
  Three 80-tone pair blocks will be used per session (~1 hour with breaks). To minimize practice effects, we will use a different base tone for each treatment day (e.g. 500, 1000, and 2000 Hz), also in a randomized counter-balanced order. To assess the improvement over a treatment day, we will record the ratio of the frequencies in all tone pairs. To correct this non-normal distribution we take the natural log of each of these ratios to determine the tone matching threshold.
Mismatch Negativity (MMN) | 3 weeks
  MMN will be obtained independently to pitch stimuli utilizing the same base frequencies as the SBR, (e.g. 500, 1000, and 2000 Hz). Two sessions will be held each day, both before and after study drug/SBR intervention. MMN will be generated using previously published methods. MMN is maximal at frontocentral electrodes (Fz, Cz). For all measures, peak amplitude at frontocentral electrodes within predefined latency range will be primary outcome measure. We primarily evaluate effect of study drug.

SECONDARY OUTCOMES:
Tone Matching | 3 weeks
  This task consists of pairs of 100-ms tones in series, with 500-ms intertone interval. Within each pair, tones are either identical or differed in frequency by specified amounts in each block (2.5%, 5%, 10%, 20%, or 50%). In each block, 12 of the tones are identical and 14 are dissimilar. Tones are derived from 3 reference frequencies (500, 1000, and 2000 Hz) to avoid learning effects.
Auditory Emotion Recognition Task | 3 weeks
  The sentences will be scored based on the speaker's intended emotion (happy, sad, angry, fear or neutral). The sentences are semantically neutral and consisted of both statements and questions (i.e., ''It is eleven o'clock'', ''Is it eleven o'clock?'').
Positive and Negative Symptom Scale (PANSS | 3 weeks
  Assesses severity of positive, negative and cognitive symptoms in SZ
Medical Symptom Inventory (aka Side Effect Checklist) | 3 weeks
  designed to assess vital signs and commonly occurring antipsychotic side effects.
MATRICS consensus cognitive battery, | 3 weeks
  Improvement is particularly expected in visual and auditory-based measures (verbal memory) as well as composite score.
Contrast sensitivity | 3 weeks
  Contrast sensitivity: stimuli consist of sine wave gratings shown side-by-side with a solid gray panel. Contrast is reduced until subjects can no longer tell the grating from the solid gray panel.
The Perceptual Organization Index (POI): | Baseline-final
  a component of the WAIS Performance IQ construct and consists of 3 tests: Picture Completion, Matrix Reasoning, and Block Design.
Emotion in motion | 3 weeks
  This is a computerized task that includes videos of faces expressing 4 basic emotions - happiness, sadness, anger, or fear - and neutral expressions.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua T Kantrowitz, MD, Principal Investigator — Columbia University/Nathan Kline Institute
Locations (1):
- Nathan Kline Insitute for Psychiatric Research, Orangeburg, New York, United States